CLINICAL TRIAL: NCT04235738
Title: Cognitive Impairment in Older Emergency Department Users and Associated Adverse Outcomes: Results From the ER2 Cohort Study Database
Brief Title: Cognitive Impairment in Older Emergency Department Users and Associated Adverse Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Professor of Geriatrics, Holder of the Dr. Joseph Kaufmann Chair in Geriatric Medicine Clinician Scientist, Department of Medicine, Division of Geriatric Medicine Director of Centre of Excellence on Longevity, RUISSS McGill, McGill University, Jewish General Hospital
Other Study IDs: 2020-2184
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Frailty; Physical Frailty; Older Emergency Department Users
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — ER2 is a simple and standardized clinical tool. The results of the questionnaires performed in ER2 study will be used. The assessment component of ER2 consists of 6 very simple closed-ended format questions (i.e., yes versus no) which are: Age category (≥ 85), male, polypharmacy (≥ 5 different medications per day), use of formal (health care or social professional) and/or informal (family and/or friend) home support, use of a walking aid regardless of its type, and temporal disorientation (inability to give the current month and/or year). A score of five points is assigned to the items "use of walking aid" and "temporal disorientation", whereas, for the other items, the assigned score is one point. The weighting of points for ER2 items is based on the results of our previous studies. Scores range from 0 (lowest risk) to 14 (highest risk). ER2 scores stratify the risk for short-term ED adverse events into three levels: low, moderate and high.

SUMMARY:
This study examines the prevalence and incidence of older ER users with cognitive impairment (i.e., dementia and/or delirium) using the ER2 item temporal disorientation in older ED users who are participants of the ER2 cohort study database.

DETAILED DESCRIPTION:
The Emergency Departments (EDs) in North America are under duress because of overcrowding, delays and diversions, which increase to epidemic proportions. The aging of Canadian's population amplifies the magnitude of this situation because older ED users are the fastest increasing group of ED users and they have complex and specific needs.

There are simple interventions with which providers must proceed in order to cure or prevent short-term ED adverse events. Delirium, motor deconditioning, polypharmacy-related adverse drug reactions, and inappropriate home support are the main conditions to target when taking care of older ED users. We previously demonstrated that acting on these conditions may significantly accelerate the discharge and significantly reduce the length of ED and hospital stay. Evidence-based medicine showed that simple and early interventions may prevent delirium (e.g., through hydration, avoiding restraint, mobilizing and satisfying basic needs, time and place reorientation) and motor deconditioning (e.g., through encouraging mobility, up to chair at mealtime during daytime hours, providing appropriate walking aid) in older patients. Medication reconciliation is also an efficient intervention to prevent adverse drug reactions. Furthermore, an early assessment of home support is a crucial step in adjusting services for an early and smooth discharge back home. Based on this evidence, we have modified the 6-item Emergency Room Evaluation and Recommendations (ER2) by adding an interventional component to the assessment portion of the tool. The interventional part depends on the assessment's results and is based on recommendations designed to encourage easy and basic interventions that prevent delirium, motor deconditioning, adverse drug interactions and inappropriate home support. These recommendations are based on answers to the ER2 items

ELIGIBILITY:
Inclusion Criteria:

- An unplanned ED visit and to be on a stretcher

Exclusion Criteria:

-

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals eligible for this study are the participants in the ER2 study.
Sampling Method: Non-Probability Sample
Enrollment: 4724 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 12 months
  The length of hospital stay is defined as the average number of days that patients spend in hospital. It will be used the ER2 tool ( Emergency Room Evaluation and Recommendation) to calculate the length of hospital stay.
Dementia | 12 months
  The diagnosis of dementia
Delirium | 12 months
  The diagnosis of delirium
Length of stay in ED | 12 months
  The length of ED stay is defined as the average number of days that patients spend in the ED. It will use the ER2 tool ( Emergency Room Evaluation and Recommendation) to calculate the length of ED stay.
Hospital admission rate | 12 months
  The number of individuals admitted to the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada